CLINICAL TRIAL: NCT07243912
Title: Evaluation of Static and Dynamic Balance, and the Effects of Joint Health, Physical Activity and Kinesiophobia on Dynamic Balance in Adult With Hemophilia.
Brief Title: Balance Evaluation in Adult Hemophilia
Status: Completed | Type: Observational
Sponsor: Ayse Merve TAT (Other)
Responsible Party: Sponsor-Investigator, Ayse Merve TAT, Assistant Professor, Yuzuncu Yil University
Organization: Yuzuncu Yil University (Other)
Other Study IDs: YuzuncuYil2025
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Postural Balance
Keywords: hemophilia; postural balance; musculoskeletal disease; physical activity; kinesiophobia
MeSH Terms: conditions — Hemophilia A; Musculoskeletal Diseases; Motor Activity; Kinesiophobia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Healthy individual
  Interventions: Diagnostic Test: Postural balance assessment
- Hemophilia Group: Adults with Hemophilia
  Interventions: Diagnostic Test: Postural balance assessment

INTERVENTIONS:
Diagnostic Test: Postural balance assessment — Static and dynamic balance was analyzed with the posturographic platform.

SUMMARY:
Introduction: Recurrent hemarthrosis in hemophilia can cause deterioration of static and dynamic balance in hemophilia. Studies in AwH report decreased dynamic balance, but consistent results regarding static balance are lacking. The causes of the decrease in dynamic balance and its associated parameters have been under explored.

Aim: To investigate static and dynamic balance in AwH compared to healthy controls and factors such as joint health, physical activity and kinesiophobia that may affect dynamic balance.

Methods: This cross-sectional controlled study included 41 AwH and 40 healthy controlled, totally 81 man and study groups determined as Hemophilia Group (HG) and Control Group (CG). Static (Static Stability Test) and dynamic balance (Limits of Stability Test (LoS) Test) were assessed Pro-kin Technobody Posturographic Platform; physical activity level with International Physical Activity Questionnaire (IPAQ) for all groups. Joint health and kinesiophobia were assessed with Hemophilia Joint Health Score and Tampa Scale for Kinesiophobia (TSK) for HG, respectively. Participants' age, height and weight were questioned in both groups, as well as type and severity of hemophilia, type of treatment, and work/job status in HG.

ELIGIBILITY:
Inclusion Criteria:

Severe or moderate hemophilia A or B

Exclusion Criteria:

Diabetus mellitus, hemiplegia, rheumatoid arthritis, Alzheimer's disease, Parkinson's disease, all vestibular system pathologies, lower extremity surgery within the last 6 months, using a walking aid.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Since hemophilia is a hereditary disease seen in males, only males were included in the control group.
Study Population: Hemophilia patients and healthy volunteers
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2025-09-10 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Static and Dynamic Balance Assessment | From enrollment to at 4 weeks
  Static and dynamic balance assessments were performed using the Pro-kin Technobody Posturographic Platform (Pro-kin 212, Technobody s.r.l., Dalmine, 21044 Bergamo, Italy). Static balance was assessed using the "Static Stability Test." This test is based on the subject's oscillations on the force platform, assessing the movement of the center of pressure, and the trunk sensor measuring trunk oscillation. Dynamic balance will be assessed using the Limits of Stability test. For the LoS test, a medium difficulty level (20 levels) will be selected from the 5-10-20-30-40 difficulty levels. Participants will be asked to orient their center of gravity toward eight directional targets for a limited time.

SECONDARY OUTCOMES:
Joint Health | From enrollment to 4 weeks
  This was assessed with Hemophilia Joint Health Score (HJHS). The HJHS evaluates the knee, elbow, and ankle index joints bilaterally and includes a walking score. Each joint can receive a maximum of 20 points, with a maximum walking score of 4 points (total score = 124). A higher score indicates poor joint health. Since the elbow joint score will not be used in this study, the maximum score was determined as 84.
Physical Activity Level | From enrollment to 4 weeks
  Physical activity was evaluated with the International Physical Activity Questionnaire (IPAQ) Short Form. The IPAQ short form consists of seven questions to be answered by the patient and asks about the duration and frequency of each activity performed during the past week. The total score is calculated in MET-min/week by multiplying the MET values defined for walking (3.3 METs), moderate-intensity physical activity (4.0 METs), and vigorous-intensity physical activity (8.0 METs) by the duration (minutes) and frequency (days). Sitting is not included in the score. High scores indicate high physical activity.
Kinesiophobia | From enrollment to 4 weeks
  Kinesiophobia will be assessed with the Tampa Scale for Kinesiophobia. Kinesiophobia is defined as the fear of reinjury and movement due to chronic pain. It consists of 17 questions, with total scores ranging 17-68. The higher the score is the gretaer the level of kinesiophobia, and scores above 37 are considered high kinesiophobia

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe M Tat, Asst Prof, Principal Investigator — Yuzuncu Yil University
Locations (1):
- Van Yüzüncü Yıl University, Van, Tuşba, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided